CLINICAL TRIAL: NCT04306211
Title: Comparison of Oxygenation Between Nasal Positive Airway Pressure (PAP) Versus Standard Care During Propofol-based Sedation for Endoscopic Ultrasound in an Ambulatory Surgical Setting: a Prospective Randomized Control Trial
Brief Title: Comparison of Oxygenation Between Nasal PAP vs Nasal During Propofol-based Sedation for EUS
Acronym: SuperNo2VA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: While there were no safety concerns, the choice of endoscopic ultrasound as part of the study design limited selection of patients. Additionally, inconsistent reliable inflation of the device was experienced during treatment.
Sponsor: Indiana University (Other)
Collaborators: Vyaire Medical (Industry)
Responsible Party: Principal Investigator, John DeWitt, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1810997768
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Endoscopic Ultrasound

STUDY DESIGN:
Intervention Model Description: Random assignment to oxygen delivery system: facial mask or SuperNO2VA Et. Crossover to other oxygen delivery system if patient experiences difficulty with assigned system.
Who Masked: Participant
Masking Description: Random assignment to oxygen delivery system: facial mask or SuperNO2VA Et. Crossover to other oxygen delivery system if patient experiences difficulty with assigned system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Facial mask (Active Comparator): facial mask for oxygen delivery
  Interventions: Device: SuperNO2VA
- SuperNO2VA (Experimental): SuperNO2VA is CPAP device to deliver oxygen with nasal mask rather than with facial mask
  Interventions: Device: SuperNO2VA

INTERVENTIONS:
Device: SuperNO2VA — SUPERNO2VA is nasal PAP device for oxygen delivery

SUMMARY:
Randomized controlled single site study involves oxygenation, continuous positive airway pressure, and ventilation of subject via nasal mask and oxygenationvia closed facemask. The intervention of the study are delivery form of supplemental oxygen, bag-mask ventilation, and continuous nasal CPAP intraoperatively and in the post anesthesia care period.

DETAILED DESCRIPTION:
124 patients with BMI> or equal to 35kg.m2 or documented Obstructive Sleep Apnea scheduled for an EUS with Propofol sedation will be randomized to CPAP vs nasal mask for oxygenation during their procedure. Patients will be monitored every 2 minutes during the procedure and in the recovery area until discharge. If patients have difficulty or refuse to wear the mask, 2 or more simultaneous or non-synchronous adverse events, change in heart rhythm or ST changes on EKG they will immediately changed to the other group. The ansethesiologist, gastroenterologist & patient will complete post-procedure questionnaires regarding their opinion of the oxygen delivery system.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or older
2. Patients undergoing upper endoscopic ultrasound
3. American Society of Anesthesiology (ASA) Physical Status I-III
4. BMI ≥35 kg/m2 or documented Obstructive Sleep Apnea
5. Has provided written informed consent

Exclusion Criteria:

1. Inpatient status
2. Active Congestive Heart Failure Exacerbation
3. Untreated ischemic heart disease
4. Acute exacerbation of respiratory disorders, including COPD and asthma
5. Emergent procedures
6. Pregnancy
7. Previous enrollment in this study
8. Inability to provide informed consent
9. Additional medical testing planned for the same day
10. History of allergic reaction to Propofol
11. Tracheostomy
12. Supra-glottic or sub-glottic tumor
13. Gastrointestinal tract obstruction or delayed transit (including delayed gastric emptying, gastric bezoar, achalasia, toxic megacolon).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M DeWitt, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Indiana University Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Facial Mask | SuperNO2VA
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Facial Mask | SuperNO2VA | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Full Range); unit: years] | 52.6 [33 to 75] | 56.17 [26 to 68] | 54.55 [26 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Benefit of Nasal PAP Versus Nasal Administration of Oxygen
Description: Compare the incidence, duration, and severity of oxygen desaturation
Time Frame: 60 minutes.
Population: Data cannot be analyzed due to unreliability. There was inadequate staff training to work the device and insufficient patients to enroll.
Arm/Group | Facial Mask | SuperNO2VA
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Total Amount of Propofol for Adequate Sedation
Description: Compares amounts of Propofol for induction and entire procedure
Time Frame: 60 minutes.
Population: as for outcome 1
Arm/Group | Facial Mask | SuperNO2VA
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Modified Observer's Assessment and Alertness/Sedation Scale (MOAAS)
Description: Compare MOAAS immediately prior to intubation and during procedure
Time Frame: 120 minutes
Population: as for outcome 1
Arm/Group | Facial Mask | SuperNO2VA
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Procedural Interruptions
Description: Compare incidence, duration and reason for procedural interruptions
Time Frame: 60 minutes
Population: as for outcome 1
Arm/Group | Facial Mask | SuperNO2VA
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 72 hours post procedure.
Arm/Group | Facial Mask | SuperNO2VA
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT04306211/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT04306211/SAP_001.pdf